CLINICAL TRIAL: NCT07185425
Title: Management of Postoperative Pain After Cesarean Delivery Using Non-pharmacological Analgesic Device, NeuroCuple™
Brief Title: Impact of the NeuroCuple Device on Pain Management After Cesarean Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: nCap Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INOVA-2025-16
Record Dates: First submitted 2025-08-29; First posted 2025-09-22 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Pain; Analgesia; Pregnancy
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Subjects who agree to participate in the study will be randomized to one of 3 groups below in a 1:1:1 allocation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and the clinical team (including obstetrics, anesthesia, operating room technicians nursing staff, and recovery and postpartum staff) will be blinded to the group assignment for the active and sham devices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- NeuroCuple device (Active Comparator): Device placed by research personnel in PACU prior to transfer to the post-partum unit
  Interventions: Device: NeuroCuple
- Sham device (Sham Comparator): Device placed by research personnel in PACU prior to transfer to the post-partum unit
  Interventions: Device: Sham
- Standard of care (No Intervention): No device will be placed

INTERVENTIONS:
Device: NeuroCuple — Device around the abdomen over c-section bandages in the PACU
  Arms: NeuroCuple device
Device: Sham — Device around the abdomen over c-section bandages in the PACU
  Arms: Sham device

SUMMARY:
This will be a single-center, sham-controlled, 3 arms, randomized (1:1:1) prospective study in females undergoing cesarean delivery to investigate the impact of NeuroCuple™ non-pharmacological analgesic device for management of postoperative pain. The investigators hypothesize that women treated with the Neurocuple device will experience less pain and consequently require less opioid pain medication after cesarean delivery compared to women who receive standard post-surgical medication.

DETAILED DESCRIPTION:
This is a single-center, sham-controlled, 3-arms, randomized, prospective study in 180 women undergoing cesarean delivery, with an expected subject enrollment duration of one year. Subjects will be screened and consented preoperatively before the scheduled case. Enrolled subjects will be randomized by research personnel using a computer generated randomization scheme in a 1:1:1 group allocation and assigned to the active device, sham device, or standard of care arms.

Upon arrival to the PACU, subjects in the standard-of-care arm will receive standard postoperative pain orders at the discretion of the primary OB/GYN. For subjects in the active and sham device arms, device will be placed as soon as feasible in the PACU and before transfer to the post-partum floor by trained research staff. Both patients and the clinical team will be blinded to the group assignment for the active and sham devices.

Pain scores will be collected from the study participants per nursing protocols while inpatient, and daily after discharge until postoperative day 4, using the Pain Numeric Rating Scale. For breakthrough pain, patients may use oral or IV opioids in the inpatient setting and oral opioids in the outpatient setting.

Upon discharge, patients are typically prescribed an opioid medication. However, this will also be left to the discretion of the primary OB/GYN. In this study, the investigators will examine total milligram morphine equivalent (MME) opioid intake at postoperative day 4 or before discharge as the primary endpoint, reduction (percentage change) in numeric pain scale as the secondary endpoint, and change in quality of recovery as the exploratory endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years or older able to provide informed consent in English or Spanish
* Scheduled for a planned or unplanned non-emergent cesarean delivery under neuraxial anesthesia
* Intact skin surfaces around the operative skin incision area at the site of patch application
* Pfannestiel skin incision

Exclusion Criteria:

* Active drug abuse
* Chronic opioid user
* Severe chronic pain
* Psoriasis vulgaris or other skin conditions precluding safe device application
* Subject is concurrently participating in another research study with an investigational drug or medical device that in the Investigator's opinion could impact subject safety or study results
* Subject with reasons to maintain an epidural beyond operative room
* Subject with complex surgery or subject who may need more than a cesarean surgery with possible tubal sterilization procedure
* Subject is deemed not suitable for the study at the discretion of the principal Investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Total Milligram Morphine Equivalents (MME) | Day of surgery to postop day 4
  Total opioid intake in MME on postoperative days 4 or before discharge.

SECONDARY OUTCOMES:
Pain reduction | Day of surgery to postop day 4
  Reduction (percentage decrease) in pain score (0-10 numeric rating scale) from day of surgery through postoperative day 4.
Quality of Recovery | Day of surgery to postop day 4
  Quality of recovery assessment evaluated on postoperative days 1-4 (Swedish Web Version of Quality of Recovery (SwQoR))
Opioid-related adverse events | Day of surgery to postop day 4
  Overall incidence of opioid-related adverse effects including maternal PONV, sedation, constipation in POD 0-4

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Saad, MD, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Fairfax Medical Campus, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Do not plan to share IPD